CLINICAL TRIAL: NCT01732497
Title: A Prospective Study of Axillary Hair Loss in Patients Treated With the miraDry System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Miramar Labs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-0009
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Underarm Hair
Keywords: Underarm Hair; Underarm Hair Reduction; Axillary Hair; Axillary Hair Reduction; Underarm Odor; Axillary Odor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Group miraDry Treatment (Experimental): This is a single group study where each enrolled subject will receive active miraDry treatment in each axilla.
  Interventions: Device: miraDry Treatment

INTERVENTIONS:
Device: miraDry Treatment — Application of electromagnetic energy to heat the lower dermis.

SUMMARY:
The purpose of this study is to evaluate hair reduction in the underarms in patients treated with the miraDry System.

DETAILED DESCRIPTION:
This study is designed to quantify the amount of hair reduction in patients treated with the miraDry System in the axilla. Hair counts will be assessed before and after treatments including at follow up visits.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Visible underarm hair (prefer light colored hair; blonde, red, gray)

Exclusion Criteria:

* Secondary Axillary Hyperhidrosis
* Prior surgery and/or Botox Injections in axillae
* Pacemaker or requires supplemental oxygen
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Patients with successful hair reduction | 3 months
  Percentage of patients that show a >=30% reduction in underarm hair at the 3 month visit compared to baseline.

SECONDARY OUTCOMES:
Patients with successful hair reduction | 12 months
  Percentage of patients that achieve a >=30% reduction in underarm hair at the 12 month visit compared to baseline

OTHER OUTCOMES:
Patient satisfaction with hair reduction | All follow-up visits through 12 months
  Patients will provide their evaluation of satisfaction with the hair reduction seen

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Quiroz, BS, RN, Study Director — Miramar Labs, Inc
Locations (3):
- United States (3):
  - Zel Skin and Laser Specialists, Edina, Minnesota
  - Laser & Skin Surgery Center of NY, New York, New York
  - Lehigh Valley Dermatology, Bethlehem, Pennsylvania

IPD SHARING:
Plan to Share IPD: No